CLINICAL TRIAL: NCT02148757
Title: Doppler Ultrasound Following Unicondylar Knee Replacement to Determine the Incidence of Postoperative DVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10093; IRB 10093 (Other Grant/Funding Number: Hospital for Special Surgeryt)
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Number of Deep Venous Thrombosis (DVT)
Keywords: DVT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DVT (Other): Doppler Ultrasound
  Interventions: Procedure: Doppler Ultrasound

INTERVENTIONS:
Procedure: Doppler Ultrasound

SUMMARY:
Purpose of this study is to determine the incidence of deep venous thrombosis after partial knee replacement.

DETAILED DESCRIPTION:
Doppler Ultrasound will be performed 2-6 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral partial knee replacement
* Postoperative anticoagulation with aspirin 325 twice daily
* Regional anesthesia
* Inflatable garments worn during hospitalization

Exclusion Criteria:

-Bilateral partial knee replacement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2011-06; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Deep venous thrombosis | 2-6 weeks after surgery

SECONDARY OUTCOMES:
body mass index | at date of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States